CLINICAL TRIAL: NCT02457845
Title: Phase I Clinical Trial of HSV G207 Alone or With a Single Radiation Dose in Children With Recurrent Supratentorial Brain Tumors
Brief Title: HSV G207 Alone or With a Single Radiation Dose in Children With Progressive or Recurrent Supratentorial Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gregory K. Friedman, MD (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Center for Advancing Translational Sciences of the National Institutes of Health (Unknown); Cannonball Kids' Cancer Foundation (Other); Rally Foundation for Childhood Cancer Research (Other); Hyundai Hope On Wheels (Other); St. Baldrick's Foundation (Other); United States Department of Defense (U.S. Federal Agency); The Andrew McDonough B+ Foundation (Other); Kaul Pediatric Research Institute (Unknown); University of Alabama at Birmingham (Other); Memorial Sloan Kettering Cancer Center (Other); Kelsie's Crew (Unknown); Eli's Block Party Childhood Cancer Foundation (Unknown); Eli Jackson Foundation (Unknown); Jaxon's F.R.O.G. Foundation (Unknown); Battle for a Cure Foundation (Unknown); Sandcastle Kids (Unknown)
Responsible Party: Sponsor-Investigator, Gregory K. Friedman, MD, Principal investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1472; R01FD005379 (FDA)
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Supratentorial Neoplasms, Malignant; Malignant Glioma; Glioblastoma; Anaplastic Astrocytoma; PNET; Cerebral Primitive Neuroectodermal Tumor; Embryonal Tumor
Keywords: Brain Tumor, Recurrent; Glioma; Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Oligodendroglioma; Rhabdoid Tumor; Cerebral Primitive Neuroectodermal Tumor; PNET; Ependymoma; Germ Cell Tumor; Choroid Plexus Carcinoma; Oncolytic Virus Therapy; Virotherapy, Oncolytic; Immunotherapy; Central Nervous System Agents; Antineoplastic Agents; Neoplasms; Pediatric; Pediatrics; Embryonal Tumor; Oncolytic; Virus; HSV; Herpes Virus
MeSH Terms: conditions — Supratentorial Neoplasms; Glioma; Glioblastoma; Astrocytoma; Neuroectodermal Tumors, Primitive; Neoplasms, Germ Cell and Embryonal; Brain Neoplasms; Gliosarcoma; Oligodendroglioma; Rhabdoid Tumor; Ependymoma; Choroid Plexus Carcinoma; Neoplasms; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSV G207 (Experimental): Single dose of HSV-1 (G207) infused through catheters into region(s) of tumor defined by MRI. If G207 is safe in the first two cohorts of patients, subsequent patients will receive a single dose of G207 infused through catheters into region(s) of tumor defined by MRI followed by a 5 Gy dose of radiation to the tumor given with 24 hours of virus inoculation.
  Intervention: Biological: G207
  Interventions: Biological: G207

INTERVENTIONS:
Biological: G207 — Single dose of HSV-1 (G207) infused through catheters into region(s) of tumor defined by MRI

SUMMARY:
This study is a clinical trial to determine the safety of injecting G207 (a new experimental virus therapy) into a recurrent or progressive brain tumor. The safety of combining G207 with a single low dose of radiation, designed to enhance virus replication and tumor cell killing, will also be tested.

DETAILED DESCRIPTION:
Outcomes for children with recurrent or progressive supratentorial malignant brain tumors are very poor, and there are a lack of effective salvage therapies once a patient fails standard treatments.

G207 is an oncolytic herpes simplex virus-1 (HSV) that has been successfully engineered to introduce mutations in the virus that enable it to selectively replicate in and kill cancer cells, but not normal cells. Replication of G207 in the tumor not only kills the infected tumor cells, but causes the tumor cell to act as a factory to produce new virus. These virus particles are released as the tumor cell dies, and can then proceed to infect other tumor cells in the vicinity, and continue the process of tumor kill. In addition to this direct oncolytic activity, the virus engenders an anti-tumor immune response; the virus is immunogenic and produces a debris field which exposes cancer cell antigens to immune cells which can target other cancer cells. Thus, the oncolytic effect of the virus and the immune response that the virus stimulates provide a one-two punch at attacking cancer cells. In preclinical studies, a single 5 Gy dose of radiation within 24 hours of virus inoculation to the tumor increased virus replication and tumor cell killing.

The University of Alabama at Birmingham has conducted three phase I trials of G207 injected into the recurrent tumor alone or combined with a single dose of radiation in adults with recurrent high-grade gliomas. In these trials, high doses (up to 3 x 10^9 plaque-forming units) of virus were safely injected directly into the tumor or surrounding brain tissue without serious toxicities. A maximum tolerated dose was not reached in all 3 trials. Radiographic and neuropathologic evidence of an antitumor response was seen in some patients. Preclinical laboratory studies have demonstrated that a variety of aggressive pediatric brain tumor types are sensitive to G207.

This study is a phase I, open-label, single institution clinical trial of G207 alone or combined with a single low dose of radiation in children with recurrent or progressive supratentorial brain tumors. The primary goal is to determine safety. The secondary aims are to obtain preliminary information on the effectiveness of and immune response to G207.

A traditional 3 + 3 design will be used with four patient cohorts. The first two cohorts will receive G207 at one of two doses, and the second two cohorts will receive G207 at one of two doses followed by a 5 Gy dose of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 36 months and < 19 years
* Pathologically proven malignant supratentorial brain tumor (including glioblastoma multiforme, giant cell glioblastoma, anaplastic astrocytoma, primitive neuroectodermal tumor, ependymoma, atypical teratoid/rhabdoid tumor, germ cell tumor, or other high-grade malignant tumor) which is progressive or recurrent despite standard care including surgery, radiotherapy, and/or chemotherapy. A pathologically proven secondary malignant tumor without curative treatment options is eligible.
* Lesion must be > 1.0 cm in diameter and surgically accessible as determined by MRI
* Patients must have fully recovered from acute treatment related toxicities of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: patients must have received their last dose at least 3 weeks prior (or at least 6 weeks if nitrosurea)
* Investigational/Biologic agents: patients must have recovered from any acute toxicities potentially related to the agent and received last dose ≥ 7 days prior to entering this study (this period must be extended beyond the time during which adverse events are known to occur for agents with known adverse events ≥ 7 days). For viral therapy, patients must have received viral therapy ≥ 3 months prior to study entry and have recovered from all acute toxicities potentially related to the agent
* Monoclonal antibodies: patient must have received last dose ≥ 21 days prior
* Radiation: Patients must have received their last fraction of craniospinal radiation (>24 Gy) or total body irradiation ≥ 3 months prior to study entry. Patients must have received focal radiation to symptomatic metastatic sites or local palliative radiation > 28 days prior to study entry.
* Autologous bone marrow transplant: Patients must be ≥ 3 months since transplant prior to study entry.
* Normal hematological, renal and liver function (Absolute neutrophil count > 1000/mm3, Platelets > 100,000/mm3, Prothrombin Time (PT) or Partial Thromboplastin Time (PTT) < 1.3 x control, Creatinine within normal institutional limits OR > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, Total Bilirubin < 1.5 mg/dl, Transaminases < 3 times above the upper limits of the institutional norm)
* Patients < 10 years, Modified Lansky score ≥ 60; patients > 10 years, Karnofsky score ≥ 60
* Patient life expectancy must be at least 8 weeks
* Written informed consent in accordance with institutional and FDA guidelines must be obtained from patient or legal guardian

Exclusion Criteria:

* Acute infection, granulocytopenia or medical condition precluding surgery
* Pregnant or lactating females
* Prior history of encephalitis, multiple sclerosis, or other central nervous system (CNS) infection
* Tumor involvement which would require ventricular, cerebellar or brainstem inoculation or would require access through a ventricle in order to deliver treatment
* Required steroid increase within 1 week prior to injection
* Known HIV seropositivity
* Concurrent therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, gancyclovir, foscarnet, cidofovir) or any immunosuppressive drug therapy (except dexamethasone or prednisone).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Measured by Frequency of Grade 3 or Above Adverse Events | Baseline to 15 years
  All events with a Grade 3 or above toxicity (defined by the CTCAE v4.0) will be tabulated by event and by relationship to G207.

SECONDARY OUTCOMES:
Immunologic Response | Baseline to 12 months
  HSV-1 antibody titers will be checked by ELISA prior to the administration of G207 and at regular intervals after treatment.
Virologic Shedding | Baseline to 15 years
  Saliva, blood and conjunctival secretions will be checked by polymerase chain reaction (PCR) and culture at regular intervals for evidence of HSV shedding and/or viremia.
Progression Free Survival | Baseline to 24 months
  Time after G207 administration to clinical and radiographic disease progression will be evaluated.
Overall Survival | Baseline to 24 months
  The overall survival for each patient receiving G207 will be calculated.
Change in Performance (Ability to Perform Normal Activities) | Baseline to 12 months
  A modified Lansky score (for children under 16 years of age) or Karnofsky score (for children 16 and older) will be recorded and measured serially with the pre-treatment score.
Quality of Life (optional) | Baseline to 12 months
  Quality of life will be measured with questionnaires taken at baseline (before administration of G207) and at specified times thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Friedman, M.D., Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (2):
- United States (2):
  - Children's of Alabama, Birmingham, Alabama
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Friedman GK, Johnston JM, Bag AK, Bernstock JD, Li R, Aban I, Kachurak K, Nan L, Kang KD, Totsch S, Schlappi C, Martin AM, Pastakia D, McNall-Knapp R, Farouk Sait S, Khakoo Y, Karajannis MA, Woodling K, Palmer JD, Osorio DS, Leonard J, Abdelbaki MS, Madan-Swain A, Atkinson TP, Whitley RJ, Fiveash JB, Markert JM, Gillespie GY. Oncolytic HSV-1 G207 Immunovirotherapy for Pediatric High-Grade Gliomas. N Engl J Med. 2021 Apr 29;384(17):1613-1622. doi: 10.1056/NEJMoa2024947. Epub 2021 Apr 10. PMID 33838625
- See also: Oncolytic HSV-1 G207 Immunovirotherapy for Pediatric High-Grade Gliomas — http://www.nejm.org/doi/full/10.1056/NEJMoa2024947

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT02457845/Prot_000.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT02457845/ICF_001.pdf